CLINICAL TRIAL: NCT01436760
Title: Genetic Contribution of Pain and Inflammation in Irritable Bowel Syndrome.
Brief Title: Genetic Contribution of Pain and Inflammation in IBS
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 132-2011
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The delinked blood/DNA is stored in the genetics laboratory and they will be analyzed for possible polymorphisms
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the study is to identify possible polymorphisms on the loci of candidate genes that may be involved in modulation of pain and inflammation in irritable bowel syndrome.

DETAILED DESCRIPTION:
Stored and de-linked blood or DNA from subjects with IBS will be utilized for analysis for possible polymorphisms at predetermined genetic loci located in chosen genes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with IBS and previously stored samples

Exclusion Criteria:

* Subjects without IBS and no previously stored samples

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Generic laboratory blood bank
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Polymorphisms | one year
  The goal of the study isd to identify possible polymorphisms on the loci of canidate genes that may be involved in modulation of pain and inflammation in irritable Bowel Syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Baharak Moshiree, MD, MS, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States